CLINICAL TRIAL: NCT03047408
Title: Evolution of REM Sleep Behavior Disorder in Parkinson's Disease Patients RBD Diagnosed Three Years Earlier
Brief Title: Evolution of RBD in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-300; 2016-A01736-45 (Other: 2016-A01736-45)
Record Dates: First submitted 2017-01-24; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: REM Sleep Behavior Disorder; Parkinson's Disease
Keywords: REM Sleep Behavior Disorder; Parkinson's Disease; REM sleep without Atonia
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with PD-RBD (Experimental): patients with PD-RBD having already underwent vPSG, clinical and neuropsychological in clinical setting or in the study "RBHP 2013 DURIF " at least three years ago.
  Interventions: Procedure: Video polysomnography

INTERVENTIONS:
Procedure: Video polysomnography — the main objective of our study is to longitudinally evaluate clinical and vPSG features of RBD, including measure of RSWA, in patients with PD-RBD, after three years from the diagnosis of RBD, in order to ascertain whether RBD features remain stable over time. The possible remission of RBD with the progression of PD would question indeed its reliability as prognostic bio-marker.

SUMMARY:
About 60% of Parkinson's Disease (PD) patients have REM sleep Behavior Disorder (RBD), a parasomnia characterized by partial or complete loss of REM sleep muscle atonia and dream-enacting behaviors, usually associated to vivid dreams. The REM Sleep without atonia is the polysomnographic hallmark of RBD, and its quantification is necessary for the diagnosis.

RBD in PD is believed to be a marker of a more widespread degenerative process and a marker of malignant phenotype. Therefore, PD patients with RBD (PD-RBD) are more severely impaired in both motor and non-motor domains, compared to those without RBD, with an increased risk of dementia. However, little is know about the relationship between the evolution of RBD, clinic and video-polysomnographic, and the progression of PD. Besides, an improvement of RBD symptoms is anecdotally reported in PD patients over time. Longitudinal evaluation of RBD in PD, assessed by questionnaires, led to controversial results, but so far, no longitudinal vPSG study has been performed in PD-RBD population.

Thus, the main objective of this study is to longitudinally evaluate clinical and video-polysomnographic features of RBD, including measure of REM Sleep without atonia, in patients with PD-RBD, after three years from the diagnosis of RBD, in order to ascertain whether RBD features remain stable over time. The possible remission of RBD with the progression of PD would question indeed its reliability as prognostic bio-marker.

DETAILED DESCRIPTION:
Type of study: longitudinal study, interventional, cross-sectional;

Number of centres: 1 (Clermont-Ferrand)

Patients: patients with Parkinson's Disease associated with REM sleep behavior disorder (PD-RBD) having already underwent video-polysomnography recording, clinical and neuropsychological evaluation in clinical setting or in the study "RBHP 2013 DURIF " at least three years ago.

Study performance:

This study will be developed in two phases:

* Phase 1 (Day 0):
* Verify inclusion criteria, receive informed and written consent;
* Demographic and clinical characteristics;
* Neurological evaluation: RBD (RBD severity scale), motor symptoms (Unified Parkinson's Disease Rating Scale, Hoeh et Yahr scale), orthostatic hypotension (Scale for outcomes in PD autonomic questionnaire), behavioral disorders hyper-dopaminergic and hypo-dopaminergic (Ardouin Scale of Behavior in Parkinson's Disease), impulsivity (Test Kirby and Stop signal reaction time)
* Dreams contents: all patients will receive 3-weeks dream diary;
* vPSG recording;
* Self-assessment questionnaires: Non-motor symptoms Questionnaire, Epworth sleepiness scale, Urgency premeditation perseverance and sensation seeking test, Aggressive questionnaire, and the Hospital Anxiety and Depression Rating Scale
* Phase 2 (+1day): Neuropsychological assessment of:
* Cognitive function, namely executive functions, visuo-spatial functions, visuo-perceptive functions (Mini mental state examination, California Verbal Learning Test, verbal fluency test, Modified Wisconsin Card Sorting Test, test de Stroop, Digit span, Visual Object and Space Perception Battery, Luria motor sequences, Rey-Osterrieth complex figure)
* Limbic functions: emotion recognition (Ekman test), apathy (Lille Apathy Rating Scale);
* Impulsivity and decision-making (Iowa Gambling test).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically confirmed idiopathic Parkinson's Disease, according to the United Kingdom Parkinson Disease Bran Bank criteria, associated with RBD, diagnosed according to the International Classification of Sleep Disorders third edition, that have been already enrolled in the study "RBHP 2013 DURIF", or that have already underwent vPSG recording,clinical and neuropsychiatric evaluation in clinical setting;
* Male and female aged between 45 to 85 years old;
* All patients are volunteers and have given written informed consent;
* All patients are able to understand and to perform all tests included in this protocol;
* User-friendly in French language, both oral and written

Exclusion Criteria:

* Patients with neurological diseases other than PD;
* Patients with psychiatric comorbidities (hallucinations, psychosis) according to the DSM-5.
* Patients with Obstructive Sleep Apnea Syndrome (Apnea/hypopnea index >15/h);
* Patients in guardianship or tutorship;
* Patients enrolled exclusively in another study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
presence of REM sleep Behavior Disorder confirmed during the video polysomnography | at day 0

SECONDARY OUTCOMES:
The REM sleep Behavior Disorder severity measured by the REM sleep Behavior Disorder scale | at day 0
The Unified Parkinson disease Rating scale score | at day 0
The behavioral disorders measured by the Ardouin Scale of Behavior in Parkinson's Disease score | at day 0
- The Orthostatic hypotension measured by the Scale for outcomes in PD- autonomic questionnaire | at day 0
The impulsivity measured by the Test of Kirby score | at day 0
The impulsivity measured by the Stop signal reaction time score | at day 0
The Hoehn and Yahr scale score | at day 0
The Non-motor symptoms Questionnaire score | at day 0
The Epworth sleepiness scale score | at day 0
The Urgency premeditation perseverance and sensation seeking test | at day 0
The Aggressive questionnaire score | at day 0
The Hospital Anxiety and Depression Rating Scale | at day 0
The dream content | at day 0
The Mini mental state examination score | at day 1
The California Verbal Learning Test score | at day 1
The fluency verbal test score | at day 1
The Modified Wisconsin Card Sorting Test | at day 1
The Stroop score | at day 1
The Empan test score | at day 1
The Visual Object and Space Perception Battery test score | at day 1
The Luria motor sequences | at day 1
The Rey-Osterrieth complex figure | at day 1
The Lille Apathy Rating Scale score | at day 1
The Iowa Gambling test score | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Livia FANTINI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France